CLINICAL TRIAL: NCT00729001
Title: Phase II, Double-blind, Randomized, Placebo-controlled Study of 2 Doses of GSK Biologicals' Live Attenuated Human Rotavirus Vaccine at Different Virus Concentrations (10 5.2 and 10 6.4 Ffu) in Healthy Infants Following a 0, 2 Month Schedule and Previously Uninfected With Human Rotavirus.
Brief Title: Study of Two Doses of GSK Biologicals' Live Attenuated HRV Vaccine (Two Different Formulations) in Healthy Infants.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 444563/005
Record Dates: First submitted 2008-08-04; First posted 2008-08-06 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Rotavirus
Keywords: Rotavirus Gastroenteritis; Human rotavirus vaccine
MeSH Terms: conditions — Rotavirus Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine; Diphtheria-Tetanus-acellular Pertussis Vaccines; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate; pentacel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Human Rotavirus Vaccine - Formulation 1
  Interventions: Biological: Human Rotavirus Vaccine - two different formulations; Biological: Prevnar; Biological: IPOL; Biological: Infanrix; Biological: OmniHIB; Biological: Pentacel
- Group B (Experimental): Human Rotavirus Vaccine - Formulation 2
  Interventions: Biological: Human Rotavirus Vaccine - two different formulations; Biological: Prevnar; Biological: IPOL; Biological: Infanrix; Biological: OmniHIB; Biological: Pentacel
- Group C (Placebo Comparator)
  Interventions: Biological: Prevnar; Biological: IPOL; Biological: Infanrix; Biological: OmniHIB; Biological: Pentacel

INTERVENTIONS:
Biological: Human Rotavirus Vaccine - two different formulations — Two oral doses
  Arms: Group A; Group B
Biological: Prevnar — Three-dose intramuscular injection (US subjects only)
Biological: IPOL — Two-dose intramuscular injection (US subjects only)
Biological: Infanrix — Three-dose intramuscular injection (US subjects only)
Biological: OmniHIB — Three-dose intramuscular injection (US subjects only)
  Other Names: ActHIB
Biological: Pentacel — Three-dose intramuscular injection (Canada only)

SUMMARY:
This is a dose exploration study to assess the safety and immunogenicity of two doses of the candidate HRV vaccine at different virus concentrations in the target age group (infants approximately 2 months of age and previously uninfected with human rotavirus) and receiving concomitant administration of routine vaccinations. The study also aims at exploring the effect of unrestricted feeding on the immunogenicity of the vaccine.

DETAILED DESCRIPTION:
All subjects enrolled from Eastern United States and Eastern Canada will continue their participation in the pilot efficacy follow-up (pilot efficacy subset).

The third dose of IPV vaccine (IPOL) may be given at visit 3, 4 or another time, at the investigator's discretion.

Comvax may be given in place of OmniHIB/ActHIB at Visit 1 and Visit 2 and the third dose of Comvax administered according to the prescribing information.

ELIGIBILITY:
Inclusion Criteria:

* A male or female child between, and including 6 and 12 weeks (42-90 days) of age at the time of the first vaccination.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Written informed consent obtained from the parents or guardians of the subject.
* Born after a normal gestation period (between 36 and 42 weeks).

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the study vaccine or placebo or planned use during the study period.
* Planned administration of a vaccine (including routine pediatric vaccines) not foreseen by the study protocol during the period starting from 14 days before each dose of vaccine(s) and ending 14 days after. Hepatitis B vaccine given concomitantly or within 14 days before and after vaccination is not an exclusion criteria.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* History of diphtheria, tetanus, pertussis, polio, Hib disease and/or invasive pneumococcal infection. History of invasive pneumococcal infection is not an exclusion criteria for Canadian subjects.
* Previous vaccination against diphtheria, tetanus, pertussis, polio, Haemophilus influenzae type b, and/or Streptococcus pneumoniae. Previous vaccination against Streptococcus pneumoniae is not an exclusion criteria for Canadian subjects.
* Use of antibiotics within 7 days preceding dose 1.
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the GI tract or other serious medical condition as determined by the investigator.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of allergic disease or reaction likely to be exacerbated by any component of the vaccine.
* Acute disease at time of enrollment.
* Gastroenteritis within 7 days preceding the study vaccine administration.
* Household contact with an immunosuppressed individual or pregnant women.
* Administration of immunoglobulins and/or blood products since birth or planned administration during the study period.
* Previous confirmed occurrence of rotavirus gastroenteritis.
* Inability to contact parents/guardians of the subject by telephone.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 529 (Actual)
Dates: Start 2000-11; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with vaccine take | Two months after the second dose
Occurrence of any grade 2 or 3 fever, vomiting or diarrhea | Within the 15-day solicited follow-up period after any dose of study vaccine.

SECONDARY OUTCOMES:
Occurrence of each type of solicited symptoms | Within the 15-day solicited follow-up period after any dose of study vaccine
Occurrence of unsolicited symptoms according to WHO classification. | Within 42 days after dose 1 and dose 2
Occurrence of serious adverse events | Throughout the entire study period
Serum rotavirus immunoglobulin A (IgA) antibody titers | At visits 1, 3 and 4 and at all Visits for pilot efficacy subset
Rotavirus seropositivity status | Before dose 1 and at the end of the study
Vaccine take (for pilot efficacy subset only) | 2 months after dose 1
Anti- polyribosyl-ribitol phosphate (PRP), anti-diphtheria and anti-tetanus toxoids, anti- pertussis toxoid (PT), anti- filamentous haemagglutinin (FHA), anti- pertactin (PRN), anti-polio type 1, 2 and 3 antibody concentrations | Two months after dose 2 and at the end of the study.
Antibody concentrations to pneumococcal serotypes 4, 6B, 9V, 14, 18C, 19F and 23F | Two months after dose 2 and at the end of the study (only in a subset of U.S. subjects)
Anti-PRP, anti-diphtheria, anti-tetanus, anti-polio type 1, 2 and 3 seroprotection status. | Two months after dose 2 and at the end of the study.
Anti-PT, anti-FHA, anti-PRN, pneumococcal serotypes 4, 6B, 9V, 14, 18C, 19F and 23F (only in US subjects) seropositivity status. | Two months after dose 2 and at the end of the study.
Seropositivity status and Geometric mean titres (GMTs) of rotavirus IgA for breast fed infants compared with formula fed infants | Two months after dose 2.
Occurrence of rotavirus gastroenteritis (in a pilot efficacy subset of subjects) | Two weeks after dose 2 until the end of the rotavirus season following vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Dennehy PH; North American Human Rotavirus Vaccine Study Group. A short report on the highlights of world-wide development of RIX4414: a North American experience comparative evaluation of safety and immunogenicity of two dosages of an oral live attenuated human rotavirus vaccine (RIX4414) in infants in the United States and Canada. Vaccine. 2006 May 1;24(18):3780-1. doi: 10.1016/j.vaccine.2005.07.030. Epub 2005 Aug 1. PMID 16111790
- [Background] Dennehy PH, Brady RC, Halperin SA, Ward RL, Alvey JC, Fischer FH Jr, Innis BL, Rathfon H, Schuind A, De Vos B; North American Human Rotavirus Vaccine Study Group. Comparative evaluation of safety and immunogenicity of two dosages of an oral live attenuated human rotavirus vaccine. Pediatr Infect Dis J. 2005 Jun;24(6):481-8. doi: 10.1097/01.inf.0000164763.55558.71. PMID 15933555
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 444563/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 444563/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 444563/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 444563/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 444563/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 444563/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register